CLINICAL TRIAL: NCT05702294
Title: A Prospective Study Looking at Improving Diagnostic Capability of Bladder Diaries by Improving Accuracy of Voided Urine Volume Measured by a Self-administered Measuring Vessel in an Ambulatory Setting in Adult Women With Lower Urinary Tract Symptoms.
Brief Title: Electronic Urinary Flowmeter to Improve Accuracy of Bladder Diaries .
Acronym: e-BLaDR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22/BW/GYN/NO/628; 296904 (Registry Identifier: IRAS ID); 22/EM/0152 (Other: REC Reference)
Record Dates: First submitted 2022-12-20; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Lower Urinary Tract Symptoms; Healthy
Keywords: electronic bladder diaries; paper bladder diaries; Overactive bladder; Urge Urinary Incontinence; Stress Urinary Incontinence; automated measurement; voided volume
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: We aim to demonstrate error in "eye-ball" (traditional method of estimating voided volumes) and increased accuracy of the automated vessel to within the internationally recognized standard of 3% using a flowmeter as the gold standard.
  We will achieve that by:
  A. Performing Bench testing. In vitro assessment to demonstrate error in "eye-ball" (traditional method of estimating voided volumes) and increased accuracy to within the internationally recognized standard of 3% using a flowmeter as the gold standard.
  B. Recruiting a control group to develop more accurate nomograms of bladder function. The control group will be blinded to the automatic cup measurements.
  C. Using the tool with women presenting to the Urogynaecology service using the conventional "eye-balling " method and automated uroflowmetry system to assess error from eye-balling and assess how the bladder diary changes comparing the two methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Adult females with no lower urinary tract symptoms will complete a 3-day paper bladder diary. After each void they will transfer their voided volume to the diary pod (vessel that calculates automatically the voided volume) for the duration of these three days.
  After three days the reports of the paper diary versus the electronic diary will be compared.
  Interventions: Device: Diary pod ( measuring vessel that automatically calculates voided volume)
- LUTS ( Lower urinary tract symptoms) arm (Experimental): Adult females with lower urinary tract symptoms will complete a 3-day paper bladder diary. After each void they will transfer their voided volume to the diary pod (vessel that calculates automatically the voided volume) for the duration of these three days.
  After three days the reports of the paper diary versus the electronic diary will be compared.
  Interventions: Device: Diary pod ( measuring vessel that automatically calculates voided volume)

INTERVENTIONS:
Device: Diary pod ( measuring vessel that automatically calculates voided volume) — Women in the control arm of the study will be required to void in the measuring cup and write down their estimates on the paper diary and then transfer the voided volume to the diary pod provided (or vice versa).
  Other Names: Minze diary pod
  Arms: Control
Device: Diary pod ( measuring vessel that automatically calculates voided volume) — Women in the Lower Urinary Tract Symptoms ( LUTS) arm of the study will be required to void in the measuring cup and write down their estimates on the paper diary and then transfer the voided volume to the diary pod provided (or vice versa).
  Other Names: Minze diary pod
  Arms: LUTS ( Lower urinary tract symptoms) arm

SUMMARY:
The goal of this clinical trial is to give an answer to the question of whether an automated calculation of voided volumes would produce a more accurate set of bladder diary data when compared to the traditional ''eye-balling'' method of estimated voided volumes of paper bladder diaries, in female adult patients with lower urinary tract symptoms (LUTS).

The main question[s] it aims to answer are:

* Does an automated measurement of voided volumes improve the accuracy of bladder diary data?
* Does an automated measurement of voided volumes improve the utility of bladder diaries?

Participants will be asked to:

* void in the disposable measuring jug and record their estimated voided volume for a total of three consecutive days in a paper diary (as per usual care).
* transfer their voided volume from the disposable jug to the automated vessel (diary pod) after each void for the same three consecutive days.

The reports generated from the paper diaries (estimated volumes) will be compared to the reports generated from the electronic automated measurement of voided volumes to understand whether there is a clinically significant difference between the two.

The investigators aim to recruit healthy female adult volunteers with no lower urinary tract symptoms to understand the normal voiding patterns and volumes of adult females using the diary pod.

The investigators will also recruit adult females with lower urinary tract symptoms and compare the two methods of capturing the voided volume

DETAILED DESCRIPTION:
Project Summary:

This study is part of a research project looking at improving accuracy and increasing the utility of bladder diaries, which form one of the most basic first line investigations in females with lower urinary tract symptoms (LUTS). It is a single centre, prospective, interventional study which will offer a vessel for automated measurement of voided volumes of urine. The accuracy of bladder diaries generated by the automated measurement will then be compared to the bladder diaries generated by the conventional eyeballing estimate method of measuring voided volumes.

The principal objective of this study is to give an answer to the question of whether an automated calculation of voided volumes would produce a more accurate set of data that would be inputted in the bladder diary of the patients and therefore improve the utility and diagnostic ability of this gold standard first line investigation.

Study Objectives (Aims):

This project aims to simplify both the collection and analysis; as a result, the test will become simpler to perform, more accurate and helpful to clinicians. It will lead to faster, more accurate assessment of LUTS in women, improving patient satisfaction whilst at the same time providing a cost-effective service.

Null hypothesis:

Automated measurement of voided volumes and improved accuracy of bladder diary data does not affect utility of bladder diaries.

Primary outcome of study:

Accuracy of measurement of voided volume with automated device (aim to be within 3%) as defined international standard.

Secondary outcome of study:

1. Outline existing evidence and identify gaps in the knowledge
2. Outline areas of future development
3. Educational purposes as it is a student research project

Methods and materials:

i. Study Design: This is a prospective, monocentric, open label, non-randomised, observational study in which the investigators aim to demonstrate error in "eye ball" (traditional method of estimating voided volumes) and increased accuracy of the automated vessel to within the internationally recognized standard of 3% using a flowmeter as the gold standard.

The investigators will achieve that by:

A. Perform Bench testing. In vitro assessment to demonstrate error in "eye-ball" (traditional method of estimating voided volumes) and increased accuracy to within the internationally recognized standard of 3% using a flowmeter as the gold standard.

B. Recruiting a control group (healthy individual adult women with no lower urinary tract symptoms) to develop more accurate nomograms of bladder function. This will require between 25-50 women of various ages. The control group will be blinded to the automatic cup measurements.

C. Using the tool with women presenting to the Urogynaecology service using the conventional "eye-balling " method and automated uroflowmetry system to assess error from eye-balling and assess how the bladder diary changes comparing the two methods. The investigators would like to recruit approximately 50 patients in each of the following groups: overactive bladder, stress incontinence and prolapse. The groups will be compared using a T test as data are normally distributed. The new nomograms will use ANOVA software and replicate the statistics already established for this. The participants in those groups will be also blinded to the automatic cup measurements generated.

D. Developing Receiver Operating characteristic (ROC) curves for potential diagnostic accuracy tests correlated with increased specificity of voided volumes for future studies.

This study design has been chosen in order to demonstrate the potential diagnostic benefits of a diary generated by an automated voiding measurement system.

Participants will be female adults who present in Urogynaecology clinics with lower urinary tract symptoms and require a bladder diary as a first line investigation tool.

Recruitment will take place in the Outpatient Urogynaecology clinic. Women presenting with lower urinary tract symptoms will be identified by the Urogynaecology team in clinic and asked to complete a 3-day paper bladder diary by voiding into the disposable paper jug (as per their usual care). For each void over the 3-day period they will be asked to transfer the voided volume from the disposable paper jug to the diary pod (automated device) which will automatically calculate the voided volume and store the result automatically to the app on their phone. The patient might choose to void first in the automated diary pod and then transfer the voided volume to the conventional paper jag. Both ways are acceptable. The participants will be blinded to those automated measurements as they will not be able to see the volume recorded on the app. All these volumes will be stored in an online electronic portal. The only person with access to the patient's portal is the clinician responsible for the research project. At the end of the 3-day period the portal will generate an automated electronic summary of the 3 day diary and this will be compared to the paper diary. The device does not require calibration as it is already pre-calibrated. A patient information leaflet will be handed out to the participants and the risks/benefits and rights to voluntarily participate and withdraw from their study explained. Informed consent will be taken in an outpatient clinic setting after the patient has read the patient information leaflet.

ELIGIBILITY:
Eligibility criteria for females with lower urinary tract symptoms:

Inclusion Criteria:

1. Females
2. 18 years of age or above
3. Females presenting with lower urinary tract symptoms

Exclusion Criteria:

1.Females who have a mental/physical disability which would make them unable to understand/comply with the requirements of the study.

Eligibility criteria for healthy volunteers:

Inclusion criteria

1. Female
2. 18 years of age or above

Exclusion criteria

1. Females who have a mental/physical disability which would make them unable to understand/comply with the requirements of the study.
2. Female with (LUTS).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-07-19 (Estimated); Study Completion 2025-07-19 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a difference of more than 3% between the estimated recorded voided volumes in milliliters (mL) and the voided volume recorded in milliliters (mL) by the automated device. | After completion of the three day bladder diary ( both paper and electronic version) of all study recruits
  We will compare the estimated volumes documented in milliliters (mL) on the paper diary by the participant versus the volumes calculated in milliliters (mL) automatically by the electronic device for each participant. We will calculate the number of participants with a difference greater than 3% between the volumes estimated in their paper bladder diary ( in mL) and the volumes measured ( in mL) automatically by their device . An error of plus or minus 3% of the voided volume in milliliters is the acceptable range as defined by the guidelines of the International Continence Society that provide a benchmark for all urodynamic equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Toozs-Hobson, MD, Principal Investigator — Birmingham Women's NHS Foundation Trust; ILIAS LIAPIS, MD, Principal Investigator — Birmingham Women's and Children's Hospital
Locations (1):
- Birmingham Women's and Children's Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No